CLINICAL TRIAL: NCT00191724
Title: Drotrecogin Alfa (Activated) (LY203638)] Exploratory, Safety Study, Multi-Center, Randomized, Placebo-Controlled, Dose Escalating Study Design, Comparing a Standard Therapy (Enoxaparin Sodium) for Submassive Pulmonary Embolism to a Combined Therapy of Drotrecogin Alfa (Activated) Plus Enoxaparin Sodium.
Brief Title: Adjuvant Treatment of Pulmonary Embolism With Drotrecogin Alfa (Activated): Phase II Exploratory Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8354; F1K-MC-O014
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2009-06-17 (Estimated); Last update posted 2009-06-24 (Estimated); Status verified 2009-06

CONDITIONS: Submassive Pulmonary Embolism
MeSH Terms: interventions — drotrecogin alfa activated; Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental)
  Interventions: Drug: Drotrecogin Alfa (Activated); Drug: Enoxaparin
- 2 (Experimental)
  Interventions: Drug: Enoxaparin; Drug: Drotrecogin Alfa (Activated)
- 3 (Experimental)
  Interventions: Drug: Enoxaparin; Drug: Drotrecogin Alfa (Activated)
- 4 (Experimental)
  Interventions: Drug: Enoxaparin; Drug: Drotrecogin Alfa (Activated)
- 5 (Placebo Comparator)
  Interventions: Drug: Enoxaparin; Drug: Placebo

INTERVENTIONS:
Drug: Drotrecogin Alfa (Activated) — 6 micrograms/kilograms/hour (ug/kg/hr), intravenous (IV), one infusion, over 12 hours
  Other Names: Xigris, LY203638
  Arms: 1
Drug: Enoxaparin — 1 milligram/kilogram (mg/kg), subcutaneous, every 12 hours until the target International Normalized Ratio (INR) is reached, minimum of 5 days
Drug: Placebo — intravenous (IV), one infusion, over 12 hours
  Arms: 5
Drug: Drotrecogin Alfa (Activated) — 12 micrograms/kilograms/hour (ug/kg/hr), intravenous (IV), one infusion, over 12 hours
  Other Names: Xigris, LY203638
  Arms: 2
Drug: Drotrecogin Alfa (Activated) — 18 micrograms/kilograms/hour (ug/kg/hr), intravenous (IV), one infusion, over 12 hours
  Other Names: Xigris, LY203638
  Arms: 3
Drug: Drotrecogin Alfa (Activated) — 24 micrograms/kilograms/hour (ug/kg/hr), intravenous (IV), one infusion, over 12 hours
  Other Names: Xigris, LY203638
  Arms: 4

SUMMARY:
An exploratory, multicenter, randomized, placebo-controlled, double blind, dose escalation study comparing a standard therapy for submassive pulmonary embolism (Enoxaparin sodium) to a combined therapy of Drotrecogin alfa (activated) plus Enoxaparin sodium.

ELIGIBILITY:
Patients with symptoms of acute pulmonary embolism (PE), without an indication for fibrinolytic therapy but with echocardiographic evidence of right ventricular dysfunction (submassive PE) within 48 hours of onset of symptoms

Inclusion Criteria:

* Clinical symptoms of Pulmonary embolism for less than 48 hours

Exclusion Criteria:

* Patients with symptoms of Pulmonary embolism for more than 48 hours

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2004-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mannheim, Germany

REFERENCES:
- [Derived] Dempfle CE, Elmas E, Link A, Suvajac N, Liebe V, Janes J, Borggrefe M. Endogenous plasma activated protein C levels and the effect of enoxaparin and drotrecogin alfa (activated) on markers of coagulation activation and fibrinolysis in pulmonary embolism. Crit Care. 2011;15(1):R23. doi: 10.1186/cc9968. Epub 2011 Jan 17. PMID 21241489
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Drotrecogin Alfa (Activated) - 6: Drotrecogin alfa (activated): 6 micrograms/kilograms/hour (ug/kg/hr) intravenous (IV), one infusion over 12 hours Enoxaparin: 1 milligram/kilogram (mg/kg), subcutaneous, every 12 hours until the target international normalized ratio (INR) is reached, minimum of 5 days
- Drotrecogin Alfa (Activated) - 12: Drotrecogin alfa (activated): 12 ug/kg/hr intravenous (IV), one infusion over 12 hours Enoxaparin: 1 mg/kg, subcutaneous, every 12 hours until the target international normalized ratio (INR) is reached, minimum of 5 days
- Drotrecogin Alfa (Activated) - 18: Drotrecogin alfa (activated): 18 ug/kg/hr intravenous (IV), one infusion over 12 hours Enoxaparin: 1 mg/kg, subcutaneous, every 12 hours until the target international normalized ratio (INR) is reached, minimum of 5 days
- Drotrecogin Alfa (Activated) - 24: Drotrecogin alfa (activated): 24 ug/kg/hr intravenous (IV), one infusion over 12 hours Enoxaparin: 1 mg/kg, subcutaneous, every 12 hours until the target international normalized ratio (INR) is reached, minimum of 5 days
- Placebo: Placebo: intravenous (IV), one infusion, over 12 hours Enoxaparin: 1 mg/kg, subcutaneous, every 12 hours until the target international normalized ratio (INR) is reached, minimum of 5 days
Period: Overall Study
Arm/Group | Drotrecogin Alfa (Activated) - 6 | Drotrecogin Alfa (Activated) - 12 | Drotrecogin Alfa (Activated) - 18 | Drotrecogin Alfa (Activated) - 24 | Placebo
Started | 6 | 9 | 9 | 8 | 15
Completed | 5 | 8 | 8 | 5 | 12
Not Completed | 1 | 1 | 1 | 3 | 3
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drotrecogin Alfa (Activated) - 6 | Drotrecogin Alfa (Activated) - 12 | Drotrecogin Alfa (Activated) - 18 | Drotrecogin Alfa (Activated) - 24 | Placebo | Total
Number analyzed (Participants) | 6 | 9 | 9 | 8 | 15 | 47
Age Continuous [Mean (Standard Deviation); unit: years] | 70.8 (4.4) | 65.7 (8.9) | 51.9 (16.5) | 45.6 (22.6) | 60.7 (21.9) | 58.7 (18.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 5 | 3 | 11 | 25
  Male | 3 | 6 | 4 | 5 | 4 | 22
Region of Enrollment [Number; unit: participants]
  Germany | 6 | 9 | 9 | 8 | 15 | 47
Medical History - Acute Coronary Syndrome/Myocardial Infarction [Number; unit: participants]
  Acute Coronary Syndrome/MI - Yes | 0 | 1 | 0 | 0 | 0 | 1
  Acute Coronary Syndrome/MI - No | 6 | 8 | 9 | 8 | 13 | 44
  Acute Coronary Syndrome/MI - Unknown | 0 | 0 | 0 | 0 | 2 | 2
Medical History - Chronic Obstructive Pulmonary Disease [Number; unit: participants]
  Chronic Obstructive Pulmonary Disease - Yes | 0 | 2 | 0 | 0 | 0 | 2
  Chronic Obstructive Pulmonary Disease - No | 5 | 7 | 9 | 8 | 13 | 42
  Chronic Obstructive Pulmonary Disease - Unknown | 1 | 0 | 0 | 0 | 2 | 3
Medical History - Deep Vein Thrombosis [Number; unit: participants]
  Deep Vein Thrombosis - Yes | 1 | 2 | 1 | 2 | 2 | 8
  Deep Vein Thrombosis - No | 2 | 7 | 8 | 6 | 13 | 36
  Deep Vein Thrombosis - Unknown | 3 | 0 | 0 | 0 | 0 | 3
Medical History - Ischemic Stroke [Number; unit: participants]
  Ischemic Stroke - Yes | 1 | 1 | 0 | 0 | 3 | 5
  Ischemic Stroke - No | 4 | 8 | 9 | 8 | 12 | 41
  Ischemic Stroke - Unknown | 1 | 0 | 0 | 0 | 0 | 1
Medical History - Pulmonary Embolism [Number; unit: participants]
  Pulmonary Embolism - Yes | 1 | 2 | 0 | 1 | 0 | 4
  Pulmonary Embolism - No | 3 | 7 | 9 | 7 | 15 | 41
  Pulmonary Embolism - Unknown | 2 | 0 | 0 | 0 | 0 | 2
Medical History - Venous Thromboembolism [Number; unit: participants]
  Venous Thromboembolism - Yes | 0 | 2 | 1 | 0 | 1 | 4
  Venous Thromboembolism - No | 3 | 7 | 8 | 7 | 12 | 37
  Venous Thromboembolism - Unknown | 3 | 0 | 0 | 1 | 2 | 6
Race/Ethnicity [Number; unit: participants]
  Caucasian | 6 | 9 | 8 | 7 | 15 | 45
  Other | 0 | 0 | 0 | 1 | 0 | 1
  Unknown | 0 | 0 | 1 | 0 | 0 | 1
Body Weight [Mean (Standard Deviation); unit: kilograms] | 76.0 (9.7) | 93.9 (13.3) | 85.2 (17.6) | 86.4 (13.8) | 85.7 (18.6) | 86.0 (16.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Bleeding Events
Description: Number of patients with major bleeding events, defined as: Reduction in hemoglobin of 2 to 5 grams per deciliter (g/dL) within 24 hours; Transfusion of 2 to 4 units of packed red blood cells within 24 hours; Hematoma requiring prolonged hospitalization or surgical intervention; Intracranial or retroperitoneal hemorrhage.
Time Frame: baseline through day 6
Population: The population analyzed was all randomized patients who received any amount of study drug [drotrecogin alfa (activated) or placebo].
Measure: Number; unit: participants
Arm/Group | Drotrecogin Alfa (Activated) - 6 | Drotrecogin Alfa (Activated) - 12 | Drotrecogin Alfa (Activated) - 18 | Drotrecogin Alfa (Activated) - 24 | Placebo
Number analyzed (Participants) | 5 | 8 | 8 | 5 | 12
participants
  Intracranial Hemorrhage | 1 | 0 | 0 | 0 | 0
  Reduction in Hemoglobin | 0 | 0 | 0 | 0 | 1
  Transfusion | 0 | 0 | 0 | 0 | 0
  Hematoma | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Right Ventricular Enddiastolic Area/Left Ventricular Enddiastolic Area (RVEDA/LVEDA) Ratios
Description: Change of right ventricular function measured as difference of right ventricular enddiastolic area/left ventricular enddiastolic area (RVEDA/LVEDA) ratios by echocardiography
Time Frame: baseline, day 6, day 90
Population: Population is all randomized patients who received any amount of study drug [drotrecogin alfa (activated) or placebo]. Patients who had no postbaseline measure at Day 6 or Day 90 were excluded from the analysis of change from baseline to day 6 or day 90, respectively.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Drotrecogin Alfa (Activated) - 6 | Drotrecogin Alfa (Activated) - 12 | Drotrecogin Alfa (Activated) - 18 | Drotrecogin Alfa (Activated) - 24 | Placebo
Number analyzed (Participants) | 6 | 9 | 9 | 8 | 15
ratio
  RVEDA/LVEDA at Day 0 | 0.8 (0.3) | 1.0 (0.3) | 1.0 (0.4) | 0.9 (0.4) | 1.1 (0.5)
  RVEDA/LVEDA at Day 6 | 0.7 (0.3) | 0.7 (0.2) | 0.8 (0.3) | 0.6 (0.2) | 0.7 (0.2)
  RVEDA/LVEDA at Day 90 | 0.5 (0.1) | 0.5 (0.1) | 0.6 (0.1) | 0.5 (0.1) | 0.6 (0.2)
Statistical Analysis 1: Comparison: Drotrecogin Alfa (Activated) - 6 vs Drotrecogin Alfa (Activated) - 12 vs Drotrecogin Alfa (Activated) - 18 vs Drotrecogin Alfa (Activated) - 24 vs Placebo; Test type: Superiority or Other; p = 0.528, Regression, Linear — P-value for effect of drotrecogin alfa (activated) dose in right ventricular function at Day 6
Statistical Analysis 2: Comparison: Drotrecogin Alfa (Activated) - 6 vs Drotrecogin Alfa (Activated) - 12 vs Drotrecogin Alfa (Activated) - 18 vs Drotrecogin Alfa (Activated) - 24 vs Placebo; Test type: Superiority or Other; p = 0.230, Regression, Linear — P-value for effect of drotrecogin alfa (activated) dose on right ventricular function at Day 90

3. Secondary Outcome: Chronic Respiratory Questionnaire Self-Administered Standardized Format (CRQ-SAS of the McMaster University Canada)
Description: Scores in each of the 4 domains (dyspnea, fatigue, emotional, and mastery) ranged from 1 (maximum impairment) to 7 (no impairment).
Time Frame: baseline and day 90 (follow-up)
Population: Population was all randomized patients who received any study drug [drotrecogin alfa (activated) or placebo]. Patients who had no postbaseline assessment were excluded from the analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drotrecogin Alfa (Activated) - 6 | Drotrecogin Alfa (Activated) - 12 | Drotrecogin Alfa (Activated) - 18 | Drotrecogin Alfa (Activated) - 24 | Placebo
Number analyzed (Participants) | 5 | 8 | 8 | 5 | 13
units on a scale
  Dyspnea - Baseline | 5.0 (1.8) | 4.5 (1.5) | 4.8 (1.6) | 5.0 (2.4) | 4.8 (1.7)
  Dyspnea - 90 Day Follow-Up | 4.8 (1.4) | 5.1 (1.7) | 6.7 (0.7) | 4.8 (2.1) | 6.5 (0.6)
  Fatigue - Baseline | 4.5 (1.5) | 3.6 (1.4) | 4.2 (1.2) | 4.7 (1.0) | 4.1 (1.3)
  Fatigue - 90 Day Follow-Up | 4.8 (1.3) | 4.1 (1.0) | 5.2 (1.1) | 4.0 (1.3) | 5.0 (0.7)
  Emotional - Baseline | 4.0 (1.2) | 4.1 (1.0) | 4.8 (1.2) | 6.1 (0.9) | 4.4 (1.1)
  Emotional - 90 Day Follow-Up | 4.7 (1.1) | 4.8 (1.3) | 5.5 (1.0) | 4.4 (1.5) | 5.2 (0.9)
  Mastery - Baseline | 5.1 (0.8) | 4.1 (1.2) | 4.7 (1.7) | 5.8 (1.4) | 4.8 (1.4)
  Mastery - 90 Day Follow-Up | 5.0 (1.2) | 4.9 (2.1) | 6.1 (1.2) | 4.9 (1.7) | 6.1 (0.9)
Statistical Analysis 1: Comparison: Drotrecogin Alfa (Activated) - 6; Test type: Superiority or Other; p = 0.018, Regression, Linear — P-value for Dyspnea 90-Day Follow-Up
Statistical Analysis 2: Comparison: Drotrecogin Alfa (Activated) - 6; Test type: Superiority or Other; p = 0.720, Regression, Linear — P-value for Emotional 90 Day Follow-up
Statistical Analysis 3: Comparison: Drotrecogin Alfa (Activated) - 6; Test type: Superiority or Other; p = 0.481, Regression, Linear — P-value for Fatigue 90 Day Follow-Up
Statistical Analysis 4: Comparison: Drotrecogin Alfa (Activated) - 6; Test type: Superiority or Other; p = 0.161, Regression, Linear — P-value for Mastery 90 Day Follow-Up
Statistical Analysis 5: Comparison: Drotrecogin Alfa (Activated) - 12; Test type: Superiority or Other; p = 0.068, Regression, Linear — P-value for Dyspnea 90 Day Follow-Up
Statistical Analysis 6: Comparison: Drotrecogin Alfa (Activated) - 12; Test type: Superiority or Other; p = 0.985, Regression, Linear — P-value for Emotional 90 Day Follow-Up
Statistical Analysis 7: Comparison: Drotrecogin Alfa (Activated) - 12; Test type: Superiority or Other; p = 0.281, Regression, Linear — P-value for Fatigue 90 Day Follow-Up
Statistical Analysis 8: Comparison: Drotrecogin Alfa (Activated) - 12; Test type: Superiority or Other; p = 0.273, Regression, Linear — P-value for Mastery 90 Day Follow-Up
Statistical Analysis 9: Comparison: Drotrecogin Alfa (Activated) - 18; Test type: Superiority or Other; p = 0.848, Regression, Linear — P-value for Dyspnea 90 Day Follow-Up
Statistical Analysis 10: Comparison: Drotrecogin Alfa (Activated) - 18; Test type: Superiority or Other; p = 0.841, Regression, Linear — P-value for Emotional 90 Day Follow-Up
Statistical Analysis 11: Comparison: Drotrecogin Alfa (Activated) - 18; Test type: Superiority or Other; p = 0.797, Regression, Linear — P-value for Fatigue 90 Day Follow-Up
Statistical Analysis 12: Comparison: Drotrecogin Alfa (Activated) - 18; Test type: Superiority or Other; p = 0.963, Regression, Linear — P-value for Mastery 90 Day Follow-Up
Statistical Analysis 13: Comparison: Drotrecogin Alfa (Activated) - 24; Test type: Superiority or Other; p = 0.149, Regression, Linear — P-value for Dyspnea 90 Day Follow-Up
Statistical Analysis 14: Comparison: Drotrecogin Alfa (Activated) - 24; Test type: Superiority or Other; p = 0.141, Regression, Linear — P-value for Emotional 90 Day Follow-Up
Statistical Analysis 15: Comparison: Drotrecogin Alfa (Activated) - 24; Test type: Superiority or Other; p = 0.774, Regression, Linear — P-value for Fatigue 90 Day Follow-Up
Statistical Analysis 16: Comparison: Drotrecogin Alfa (Activated) - 24; Test type: Superiority or Other; p = 0.394, Regression, Linear — P-value for Mastery 90 Day Follow-Up

4. Secondary Outcome: Difference in Pulmonary Artery (PA) Pressure
Description: Investigator decided estimate of pulmonary artery pressure by echocardiography would not be useful and no data on pulmonary artery pressure were collected.
Time Frame: baseline, day 6, day 90
Population: Data were not collected.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Drotrecogin Alfa (Activated) - 6 | Drotrecogin Alfa (Activated) - 12 | Drotrecogin Alfa (Activated) - 18 | Drotrecogin Alfa (Activated) - 24 | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Drotrecogin Alfa (Activated) - 6 | Drotrecogin Alfa (Activated) - 12 | Drotrecogin Alfa (Activated) - 18 | Drotrecogin Alfa (Activated) - 24 | Placebo
Serious Adverse Events (participants affected / at risk) | 1 | 1 | 1 | 2 | 2
Other Adverse Events (participants affected / at risk) | 3 | 8 | 8 | 6 | 11
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Drotrecogin Alfa (Activated) - 6 | Drotrecogin Alfa (Activated) - 12 | Drotrecogin Alfa (Activated) - 18 | Drotrecogin Alfa (Activated) - 24 | Placebo
Abdominal pain (Gastrointestinal disorders) | 0/6 (0) | 1/9 (1) | 0/9 (0) | 0/8 (0) | 0/15 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 1/15 (1)
Atrial flutter (Cardiac disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 1/15 (1)
Bradycardia (Cardiac disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 1/15 (1)
Cardiac arrest (Cardiac disorders) | 0/6 (0) | 0/9 (0) | 1/9 (1) | 0/8 (0) | 0/15 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 1/9 (1) | 0/9 (0) | 0/8 (0) | 0/15 (0)
Deep vein thrombosis (Vascular disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 1/8 (1) | 0/15 (0)
Oedema peripheral (General disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 1/8 (1) | 0/15 (0)
Prothrombin time prolonged (Investigations) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 1/15 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 1/8 (1) | 0/15 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 0/9 (0) | 1/9 (1) | 0/8 (0) | 0/15 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1/6 (1) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 0/15 (0)
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Drotrecogin Alfa (Activated) - 6 | Drotrecogin Alfa (Activated) - 12 | Drotrecogin Alfa (Activated) - 18 | Drotrecogin Alfa (Activated) - 24 | Placebo
Splenomegaly (Blood and lymphatic system disorders) | 0/6 (0) | 0/9 (0) | 1/9 (1) | 1/8 (1) | 0/15 (0)
Palpitations (Cardiac disorders) | 0/6 (0) | 0/9 (0) | 2/9 (2) | 0/8 (0) | 0/15 (0)
Tachycardia (Cardiac disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 1/8 (1) | 0/15 (0)
Vertigo (Ear and labyrinth disorders) | 0/6 (0) | 0/9 (0) | 2/9 (2) | 1/8 (1) | 2/15 (2)
Abdominal pain (Gastrointestinal disorders) | 0/6 (0) | 1/9 (1) | 0/9 (0) | 0/8 (0) | 0/15 (0)
Colonic polyp (Gastrointestinal disorders) | 0/6 (0) | 1/9 (1) | 0/9 (0) | 0/8 (0) | 0/15 (0)
Diarrhoea (Gastrointestinal disorders) | 0/6 (0) | 0/9 (0) | 1/9 (1) | 1/8 (1) | 1/15 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 1/15 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 1/15 (1)
Dyspepsia (Gastrointestinal disorders) | 0/6 (0) | 1/9 (1) | 1/9 (1) | 0/8 (0) | 1/15 (1)
Gastritis (Gastrointestinal disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 1/8 (1) | 1/15 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1/6 (1) | 1/9 (1) | 0/9 (0) | 0/8 (0) | 0/15 (0)
Haemorrhoids (Gastrointestinal disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 1/15 (2)
Hiatus hernia (Gastrointestinal disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 2/8 (2) | 2/15 (2)
Intestinal perforation (Gastrointestinal disorders) | 0/6 (0) | 1/9 (1) | 0/9 (0) | 0/8 (0) | 0/15 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0/6 (0) | 0/9 (0) | 1/9 (1) | 0/8 (0) | 1/15 (1)
Nausea (Gastrointestinal disorders) | 0/6 (0) | 0/9 (0) | 3/9 (3) | 0/8 (0) | 1/15 (1)
Reflux oesophagitis (Gastrointestinal disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 1/8 (1) | 0/15 (0)
Vomiting (Gastrointestinal disorders) | 0/6 (0) | 0/9 (0) | 2/9 (2) | 0/8 (0) | 0/15 (0)
Catheter site oedema (General disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 1/15 (1)
Catheter site pain (General disorders) | 0/6 (0) | 0/9 (0) | 1/9 (1) | 0/8 (0) | 0/15 (0)
Catheter site related reaction (General disorders) | 0/6 (0) | 0/9 (0) | 1/9 (1) | 0/8 (0) | 0/15 (0)
Chest pain (General disorders) | 0/6 (0) | 0/9 (0) | 2/9 (2) | 0/8 (0) | 0/15 (0)
Discomfort (General disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 1/8 (1) | 0/15 (0)
Fatigue (General disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 2/8 (2) | 0/15 (0)
Inflammation (General disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 1/8 (1) | 0/15 (0)
Injection site haemorrhage (General disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 1/8 (1) | 0/15 (0)
Oedema peripheral (General disorders) | 0/6 (0) | 1/9 (1) | 0/9 (0) | 2/8 (3) | 0/15 (0)
Polyp (General disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 1/15 (1)
Vessel puncture site haematoma (General disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 1/15 (1)
Pyrexia (General disorders) | 0/6 (0) | 1/9 (1) | 3/9 (3) | 0/8 (0) | 0/15 (0)
Hepatic cyst (Hepatobiliary disorders) | 0/6 (0) | 0/9 (0) | 1/9 (1) | 0/8 (0) | 1/15 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0/6 (0) | 0/9 (0) | 2/9 (2) | 1/8 (1) | 1/15 (1)
Hepatomegaly (Hepatobiliary disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 1/15 (1)
Portal hypertensive gastropathy (Hepatobiliary disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 1/8 (1) | 0/15 (0)
Drug hypersensitivity (Immune system disorders) | 0/6 (0) | 0/9 (0) | 1/9 (1) | 0/8 (0) | 0/15 (0)
Bronchitis (Infections and infestations) | 0/6 (0) | 0/9 (0) | 1/9 (1) | 0/8 (0) | 0/15 (0)
Clostridium difficile colitis (Infections and infestations) | 0/6 (0) | 1/9 (1) | 0/9 (0) | 0/8 (0) | 0/15 (0)
Cystitis (Infections and infestations) | 0/6 (0) | 1/9 (1) | 0/9 (0) | 0/8 (0) | 1/15 (1)
Eye infection (Infections and infestations) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 1/15 (1)
Influenza (Infections and infestations) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 1/15 (1)
Nasopharyngitis (Infections and infestations) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 1/8 (1) | 0/15 (0)
Pneumonia (Infections and infestations) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 1/15 (1)
Pyelonephritis (Infections and infestations) | 0/6 (0) | 0/9 (0) | 1/9 (1) | 0/8 (0) | 0/15 (0)
Urethritis (Infections and infestations) | 0/6 (0) | 0/9 (0) | 1/9 (1) | 0/8 (0) | 0/15 (0)
Overdose (Injury, poisoning and procedural complications) | 0/6 (0) | 1/9 (1) | 0/9 (0) | 0/8 (0) | 0/15 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1/6 (1) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 0/15 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1/6 (1) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 0/15 (0)
C-reactive protein increased (Investigations) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 1/8 (1) | 0/15 (0)
Haemoglobin decreased (Investigations) | 1/6 (1) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 1/15 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/6 (0) | 1/9 (1) | 1/9 (1) | 0/8 (0) | 0/15 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0/6 (0) | 1/9 (1) | 0/9 (0) | 0/8 (0) | 0/15 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0/6 (0) | 1/9 (1) | 1/9 (1) | 0/8 (0) | 0/15 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0/6 (0) | 0/9 (0) | 1/9 (2) | 0/8 (0) | 0/15 (0)
Akathisia (Nervous system disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 1/15 (1)
Dementia (Nervous system disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 1/15 (1)
Headache (Nervous system disorders) | 0/6 (0) | 0/9 (0) | 1/9 (1) | 0/8 (0) | 1/15 (1)
Migraine (Nervous system disorders) | 0/6 (0) | 1/9 (2) | 0/9 (0) | 0/8 (0) | 0/15 (0)
Neuropathy peripheral (Nervous system disorders) | 0/6 (0) | 0/9 (0) | 1/9 (1) | 0/8 (0) | 0/15 (0)
Partial seizures (Nervous system disorders) | 1/6 (1) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 0/15 (0)
Presyncope (Nervous system disorders) | 0/6 (0) | 0/9 (0) | 1/9 (1) | 0/8 (0) | 0/15 (0)
Agoraphobia (Psychiatric disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 1/8 (1) | 0/15 (0)
Confusional state (Psychiatric disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 1/8 (1) | 0/15 (0)
Insomnia (Psychiatric disorders) | 1/6 (1) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 0/15 (0)
Oliguria (Renal and urinary disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 1/15 (1)
Renal cyst (Renal and urinary disorders) | 0/6 (0) | 0/9 (0) | 1/9 (1) | 0/8 (0) | 1/15 (2)
Renal pain (Renal and urinary disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 1/15 (1)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0/6 (0) | 0/9 (0) | 1/9 (1) | 0/8 (0) | 0/15 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0/6 (0) | 0/9 (0) | 1/9 (1) | 0/8 (0) | 0/15 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 1/15 (1)
Dsypnoea (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 0/9 (0) | 1/9 (1) | 0/8 (0) | 1/15 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 1/9 (1) | 1/9 (1) | 0/8 (0) | 1/15 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 0/9 (0) | 1/9 (1) | 1/8 (1) | 0/15 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 1/9 (1) | 0/9 (0) | 0/8 (0) | 0/15 (0)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 0/9 (0) | 1/9 (1) | 0/8 (0) | 0/15 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 0/9 (0) | 1/9 (1) | 0/8 (0) | 0/15 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 0/9 (0) | 1/9 (1) | 0/8 (0) | 0/15 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 1/15 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 0/9 (0) | 1/9 (1) | 0/8 (0) | 0/15 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 1/8 (1) | 0/15 (0)
Acne (Skin and subcutaneous tissue disorders) | 0/6 (0) | 0/9 (0) | 1/9 (1) | 0/8 (0) | 0/15 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0/6 (0) | 1/9 (1) | 0/9 (0) | 0/8 (0) | 0/15 (0)
Rash (Skin and subcutaneous tissue disorders) | 0/6 (0) | 0/9 (0) | 1/9 (2) | 0/8 (0) | 0/15 (0)
Angiodysplasia (Vascular disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 1/15 (1)
Haematoma (Vascular disorders) | 0/6 (0) | 0/9 (0) | 1/9 (1) | 0/8 (0) | 0/15 (0)
Hypertension (Vascular disorders) | 0/6 (0) | 1/9 (1) | 1/9 (1) | 1/8 (1) | 0/15 (0)
Phlebitis (Vascular disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 1/15 (1)
Vasodilatation (Vascular disorders) | 0/6 (0) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 1/15 (1)

LIMITATIONS AND CAVEATS:
This study was stopped early after 47 patients had been enrolled (planned enrollment was 48 patients). Study was stopped early due to slow enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days